CLINICAL TRIAL: NCT04740606
Title: A Real World Case Registry Study to Evaluate Augmented Reality Navigation System for Diagnosis of Peripheral Pulmonary Nodules
Brief Title: Airway Navigation Database Asia for Diagnosis of Peripheral Pulmonary Nodules
Acronym: ANDA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Hong Kong Sanatorium & Hospital (Industry); Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, ShiYue Li, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: 20201222
Record Dates: First submitted 2021-02-04; First posted 2021-02-05 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Lung; Node
Keywords: Augmented Reality Navigation System; Peripheral Pulmonary Nodules; biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment Group: The patients whose chest CT images show that the pulmonary nodules are highly suspected of malignant and scheduled to be diagnosed by bronchoscopy under the guidance of the Augmented Reality Navigation System.
  Interventions: Device: Augmented Reality Navigation System

INTERVENTIONS:
Device: Augmented Reality Navigation System — Investigators will assess the nodules based on the CT images of subjects before procedure. And then, the appropriate intra-airway path planned by the Augmented Reality Navigation System will be selected. The bronchoscopy with intra-airway navigation under the guidance of the Augmented Reality Navigation System will be performed and the following surgical information will be record.

SUMMARY:
The study is designed to evaluate the efficacy and safety of Augmented Reality Navigation System through intra-airway navigation system to guide bronchoscopy in the diagnosis of peripheral pulmonary nodules and explore the factors of diagnosis yield.

DETAILED DESCRIPTION:
This is a single-arm, prospective, Asian multicenter, Real World case Registry study. Recruitment is expected to last up to 12 months, and each subject may be followed up for 12 months at most after surgery which depends on certain factors. The total duration of the study is about 24 months.The research is planned to be carried out at more than 10 sites.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18;
2. Chest thin-layer CT show that the peripheral pulmonary nodule (maximum diameter ≤3 cm) is not clearly diagnosed, and planned to be sampled and diagnosed by Augmented Reality Navigation System guided bronchoscopy;
3. The target nodule is evaluated as being able to be reached via bronchoscope under the guidance of Augmented Reality Navigation System before procedure;
4. Patients can understand the study and sign informed consent form.

Exclusion Criteria:

-

1. Contraindications for bronchoscopy:

1. Myocardial infarction whithin 1 month.
2. Active massive hemoptysis.
3. Coagulation dysfunction.
4. Pregnancy.
5. Malignant arrhythmia, severe cardiac insufficiency, extreme systemic failure, etc.

2. Severe cardiopulmonary dysfunction and other diseases that may significantly increase the risk of procedure; 3. The situations in which the investigators consider that patients are not suitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients expected to be enrolled in this study is those whose chest CT images show the pulmonary nodules are highly suspected of malignant and scheduled to be diagnosed by bronchoscopy under the guidance of the Augmented Reality Navigation System.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-10 (Estimated); Primary Completion 2023-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | twelve months
  It is defined as the percentage of patients who get definitive diagnosis via bronchoscope biopsy guided by intra-airway navigation system.

SECONDARY OUTCOMES:
Diagnostic yield | Twelve months
  It is defined as the percentage of patients who get definitive diagnosis via bronchoscope biopsy guided by intra-airway navigation system.
Success rate of biopsy | Immediately after Each Operation
  It is defined as the percentage of nodules with successful biopsy.
Navigation success rate | Immediately after Each Operation
  It is defined as the percentage of nodules whose arrival is confirmed by endobronchial ultrasound (and/or fluoroscopy, or direct bronchoscopy).
Total navigation time | Immediately after Each Operation
  It is defined as the total time from the beginning of navigation to the end of navigation.
Bronchoscope operation time | Immediately after each operation
  It is defined as the total time of bronchoscope insertion to bronchoscope withdrawal.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Diseases, Guangzhou, Guangdong, China